CLINICAL TRIAL: NCT00129649
Title: Service Development: Assessing Non-attendance Rates in Outpatient Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NHLICX3806
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Asthma; Sleep Apnea Syndromes; Tuberculosis; COPD
Keywords: Telephone reminder
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes; Tuberculosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): This group received usual care and did not receive a telephone reminder
- telephone reminder group (Active Comparator): This group received a telephone reminder for their clinic appointment
  Interventions: Behavioral: Telephone reminder call

INTERVENTIONS:
Behavioral: Telephone reminder call
  Arms: telephone reminder group

SUMMARY:
Many studies have shown a high non-attendance rate in hospital outpatient clinics. The investigators have found a non-attendance rate of 25% in their asthma clinics and would like to investigate whether a reminder phone call will improve attendance rates. Patients will be randomised into two groups; one group will receive a reminder phone call one week prior to their hospital consultation and the other group will be managed in the standard manner (i.e. no reminder of any sort). The phone calls will be carried out on a Friday afternoon by a respiratory nurse specialist and a research officer for two asthma clinics based on a Wednesday morning and a Thursday afternoon.

DETAILED DESCRIPTION:
Many studies have shown a high non-attendance rate in hospital outpatient clinics. The investigators have found a non-attendance rate of 25% in their asthma clinics and would like to investigate whether a reminder phone call will improve attendance rates. Patients will be randomised into two groups; one group will receive a reminder phone call one week prior to their hospital consultation and the other group will be managed in the standard manner (i.e. no reminder of any sort). The phone calls will be carried out on a Friday afternoon by a respiratory nurse specialist and a research officer for two asthma clinics based on a Wednesday morning and a Thursday afternoon.

To have an 80% chance of detecting a 10% reduction in non-attendance rates (at 5%) 500 patients are required for this study. The rate of non-attendance will be monitored for all the patients in both groups and some demographic information will be recorded for each patient(age, sex, diagnosis and home postcode).

ELIGIBILITY:
Inclusion Criteria:

* Patients with appointments booked for 2 respiratory outpatient clinics

Exclusion criteria

Patients likely to only need one appointment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martyn R Partridge, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- NHLI Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts N, Meade K, Partridge M. The effect of telephone reminders on attendance in respiratory outpatient clinics. J Health Serv Res Policy. 2007 Apr;12(2):69-72. doi: 10.1258/135581907780279567. PMID 17407654

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone Reminder Group: This group received a telephone reminder for their clinic appointment
  Telephone reminder call
Period: Overall Study
Arm/Group | Control Group | Telephone Reminder Group
Started | 258 | 246
Completed | 182 | 181
Not Completed | 76 | 65
Not completed — Withdrawal by Subject | 76 | 65

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Telephone Reminder Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized
Sex/Gender, Customized
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Attendance Rates at Respiratory Outpatient Clinics
Description: rates of attendance measured for scheduled clinics - attended patients
Time Frame: after phone call within 1 week
Population: Lower participants number in the telephone reminder group, only participants who were could be contacted before the appointment
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Telephone Reminder Group
Number analyzed (Participants) | 258 | 104
Participants | 183 | 89
Statistical Analysis 1: Comparison: Control Group vs Telephone Reminder Group; Test type: Superiority; p = 0.004, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Control Group | Telephone Reminder Group
All-Cause Mortality (participants affected / at risk) | 0/258 | 0/246
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/246
Other Adverse Events (participants affected / at risk) | 0/258 | 0/246

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes